CLINICAL TRIAL: NCT02486770
Title: A Phase 1 Single-center (U.S.), Open Label, Dose-escalation Study of the Safety and Pharmacokinetics of Single Doses of Intravenous AerucinTM in Healthy Adult Subjects
Brief Title: Study of Single Doses of IV Aerucin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ARC-11-01
Record Dates: First submitted 2015-04-08; First posted 2015-07-01 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Aerucin 2.0mg/kg
  Interventions: Biological: Aerucin 2.0mg/kg
- Group 2 (Experimental): Aerucin 8.0mg/kg
  Interventions: Biological: Aerucin 8.0mg/kg
- Group 3 (Experimental): Aerucin 20.0mg/kg
  Interventions: Biological: Aerucin 20.0 mg/kg

INTERVENTIONS:
Biological: Aerucin 2.0mg/kg — IV Aerucin 2.0 mg/kg over 1 hour
  Arms: Group 1
Biological: Aerucin 8.0mg/kg — IV Aerucin 8.0 mg/kg over 1 hour
  Arms: Group 2
Biological: Aerucin 20.0 mg/kg — IV Aerucin 20 mg/kg over 1 hour
  Arms: Group 3

SUMMARY:
This study will evaluate the safety profile and pharmacokinetic behavior of a single administration of Aerucin in healthy adults at three different dosages.

DETAILED DESCRIPTION:
This Phase I trial will be conducted as an open label trial in 15 healthy adults. All subjects will receive a specific intravenous dose of Aerucin. There are three study groups, each with a specific dose of Aerucin. Study Group 1 will receive 2.0 mg/ kg of Aerucin . Study Group 2 will receive 8.0 mg/kg of Aerucin . Study Group 3 will receive 20 mg/kg of Aerucin . The dose levels of Aerucin are selected for this study based on animal studies showing protection in an animal model and absence of adverse effects in toxicological studies. Groups will be enrolled sequentially.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent process
2. Is male or female
3. Is age ≥18 years and ≤50 years
4. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
5. Agrees to avoid elective surgery for the duration of the study
6. For female subjects: agrees to have avoided pregnancy from 14 days prior to Study Day 0 through the duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include: a sterile sexual partner; sexual abstinence (not engaging in any sexual intercourse); hormonal contraceptives (oral, injection, transdermal patch, or implant); vaginal ring; intrauterine device (IUD); or condom.
7. Has general good health, confirmed by medical history and physical examination
8. Has body mass index (BMI) between 18 and 30 (weight/height) -

Exclusion Criteria:

1. Oral temperature ≥37.5°C
2. Abnormal CBC laboratory values (per local laboratory parameters) from blood collected at screening (>5% above ULN or >5% below LLN)
3. Abnormally elevated laboratory values (per local laboratory parameters) from blood collected at screening for ALT, AST, total bilirubin, alkaline phosphatase (ALP), blood urea nitrogen (BUN), creatinine (Cr), (>10% above ULN)
4. Abnormal urinalysis that, in the opinion of the investigator, is clinically significant
5. Positive screening urine test for illicit drugs (opiates, cocaine, amphetamines)
6. Has received an immunoglobulin product in the 120 days prior to Study Day 0
7. History or evidence of autoimmune disease
8. History or evidence of any past, present, or future possible immunodeficiency state, including laboratory evidence of HIV 1 infection.
9. History or evidence of chronic hepatitis
10. History of evidence of Pseudomonas infection
11. Received a systemic antibiotic with 14 days prior to Study Day 0
12. Participation in any other investigational study during the study period
13. Received immunoglobulin or blood products within 90 days prior to Study Day 0
14. Received any investigational drug therapy or investigational drug within 60 days prior to Study Day 0
15. Received immunosuppressive medications other than inhaled or topical immunosuppressants within 45 days prior to Study Day 0
16. Inability to discontinue daily medications during the study other than: oral contraceptives, vitamins, nonprescription nutritional supplements, aspirin, antihistamines inhaled corticosteroids, inhaled beta agonists, inhaled anticholinergics
17. All female subjects: currently pregnant or lactating/nursing; positive screening urine pregnancy test; or positive urine pregnancy test on the day of any study dosing
18. History or evidence of allergic disease or reaction that, in the opinion of the investigator, may compromise the safety of the subject
19. History or evidence of any other acute or chronic disease that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the drug or compromise the safety of the subject
20. Medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol
21. Any other reason at discretion of the investigator -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 and 84 days following dosing
  Number and % of subjects experiencing adverse events following dosing
Serious Adverse Events | 24 and 84 days following dosing
  Number and % of subjects experiencing Serious Adverse Events following dosing
Solicited Adverse Events | 7 days following dosing
  Number and % of subjects experiencing Solicited Adverse Events following dosing

SECONDARY OUTCOMES:
CMax -Observed maximum plasma concentration | 84 days following dosing
  Pharmacokinetics Characteristics
TMax-Time to reach maximum plasma concentration | 84 days following dosing
  Pharmacokinetics Characteristics
AUC0-last Area under the the concentration time curve | 84 days following dosing
  Pharmacokinetics Characteristics
AUC0-∞ Area under the concentration time curve from zero to infinite time | 84 days following dosing
  Pharmacokinetics Characteristics
Terminal phase elimination rate | 84 days following dosing
  Pharmacokinetics Characteristics
Terminal elimination half-life | 84 days following dosing
  Pharmacokinetics Characteristics

OTHER OUTCOMES:
Anti-Aerucin Antibodies | 84 days following dosing
  Exploratory analysis-evaluation of development of antibodies may be performed

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al-Ibrahim, MD, Principal Investigator — SNBL
Locations (1):
- SNBL-CPC, Baltimore, Maryland, United States